CLINICAL TRIAL: NCT01563822
Title: Phase I Study of the Effect of Flushing the Uterine Cavity With Follicular Fluid After Ovum Pick-up on Implantation Rates in ICSI Cycles
Brief Title: Does Flushing the Uterine Cavity With Follicular Fluid After Ovum Pick-up Improve Implantation Rates in ICSI Cycles?
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nawara Mohamed Hashish (Other)
Responsible Party: Sponsor-Investigator, Nawara Mohamed Hashish, Assistant professor of Obstetrics and Gynecology, Kasr El Aini Hospital
Organization: Kasr El Aini Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 132012
Record Dates: First submitted 2012-03-20; First posted 2012-03-27 (Estimated); Last update posted 2012-10-10 (Estimated); Status verified 2012-10

CONDITIONS: Intra-cytoplasmic Sperm Injection Outcome
Keywords: Follicular Fluid; uterine cavity; Implantation rates; ICSI

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- follicular fluid group (Experimental): Follicular fluid group is the group in which flushing of the uterine cavity with follicular fluid after ovum pick-up is done.
  Interventions: Biological: Follicular fluid
- control group (No Intervention): Control group is the group in which flushing of the uterine cavity with follicular fluid after ovum pick-up is not done.

INTERVENTIONS:
Biological: Follicular fluid — The intervention is flushing the uterine cavity with 2 ml of clear follicular fluid surrounding mature oocytes after ovum pick-up through an IUI catheter
  Arms: follicular fluid group

SUMMARY:
Background:

Traditionally during ovum pick-up in ICSI, we aspirate the follicles for oocyte retrieval but unfortunately we don't make use of the follicular fluid (FF) and we discard it in spite of the fact that this does not happen in nature. The fallopian tube picks-up the FF with the oocyte during ovulation. As this fluid contains stem cell factor and C-Kit receptor responsible for implantation and IGF responsible for endometrial growth and TGF that improves implantation. That's why flushing the endometrial cavity with FF after ovum pick-up might improve endometrial receptivity and implantation rates; the limiting step in ICSI.

Patients and Methods:

100 patients attending kasr El-Aini IVF center preparing for ICSI cycles are randomized into two groups. In the study group, flushing the endometrial cavity with 2ml of clear follicular fluid surrounding mature oocytes through an IUI catheter is done after ovum pick-up While in the control group, no flushing of the endometrial cavity with FF is done. The implantation rates and pregnancy rates in both groups will be assessed.

DETAILED DESCRIPTION:
Introduction:

Looking at the process of IVF, we found that we only make use of the ovum and sperm and we neglect completely the valuable effect of the follicular fluid which is currently attracting a lot of attention. Several studies revealed a pivotal role played by this fluid in the process of fertilization and implantation as it is rich in growth factors as stem cell factor, transforming growth factor and insulin growth factor and cytokines (1,2).

Macciò study confirmed that follicular fluid (FF) contains factors that induce immunosuppression and explained that the immunosuppressive activity of FF is mediated by the specific inhibition of the production of IL-1 alpha and IL-2 and by the decreased expression of the CD25 (3).

During ovum pick-up, we aspirate all the FF and throw it away after ovum retrieval. This fluid normally enters the fallopian tubes while picking the ovum during ovulation in natural cycles and it reaches the uterine cavity as well and several studies suggested that it might have a crucial role in modifying uterine receptivity preparing the endometrium for the fertilized ovum arriving after 3 days as the TGF controls apoptosis, the IGF improves endometrial thickness and the immunosuppressive activity of the FF paves the way for the embryo to implant in the uterine cavity (4,5).

Actually Hunter study in 2007, provided circumstantial evidence for entry of follicular fluid into the Fallopian tubes, especially close to the time of ovulation, with the suggestion that such entry could modify the nature of endosalpingeal secretion and transudation. Thereafter, the spectrum of gonadal hormones in follicular fluid could be influencing uterine tissues in a local manner (5).

At the same time, it is a well known fact that implantation is the limiting step in IVF success , actually almost all IVF cycles succeed in offering fertilized ova giving rise to embryos at the different stages of development but unfortunately when we transfer them to the uterine cavity, 60% fail to implant.

Implantation is a complex initial step in the establishment of a successful pregnancy. Although embryo quality is an important determinant of implantation, temporally co-ordinated differentiation of endometrial cells to attain uterine receptivity and a synchronized dialogue between maternal and embryonic tissues are crucial. Optimizing endometrial receptivity in fertility treatment will improve success rate.

Several growth factors and cytokines appear to be involved in the process of implantation. Stem cell factor and its receptor c-kit regulate the progression and survival of germ cells and play an important role in follicular development. It is present in the follicular fluid however little information was available on the role of stem cell factor and its receptor in the process of blastocyst implantation. It was not until Mitsunari examined the expression of stem cell factor and its receptor in mouse embryos and in the stromal and epithelial cells of the uterine endometrium by reverse transcription -polymerase chain reaction . He illustrated that stem cell factor derived from endometrial cells and the implanting embryo exerts paracrine and autocrine action on the process of implantation by stimulating trophoblast outgrowth through its receptor c-kit (6).

Neglecting the importance of the follicular fluid and throwing it away during the process of IVF is actually a deviation from what happens in nature where the fallopian tube is intelligent enough to appreciate the value of this fluid and pick it up with the ovum.

That is why in this study, we want to mimic natural cycles and explore the benefits of flushing the uterine cavity with follicular fluid after ovum pick-up in improving implantation rates in ICSI cycles.

Materials and methods:

100 patients attending kasr El-Ainey IVF center preparing for ICSI cycles will be randomized into two groups.

In this prospective interventional study, the patients of both groups will receive the same induction protocol for controlled ovarian hyperstimulation which is the long protocol, our standard protocol in the center. Initial suppression of ovarian function with gonadotrophin releasing hormone agonist will start on day 21 of the preceeding cycle. Human menopausal gonadotrophin induction will start after confirmed ovarian down regulation by both laboratory investigations and ultrasound by daily intramuscular injection of 150-300 IU (Merional, IBSA) until at least 3 follicles reach 18 mm and serum estradiol level lies between 1000-4000 then 10000 IU, HCG is given.

Ovum pick-up is scheduled 35 hours later, where each follicle is aspirated in a separate tube and will be examined by the embryologist separately where:

* The follicular fluid from empty follicles will be discarded, only the FF from follicles where mature oocytes were retrieved will be used.
* The follicular fluid contaminated with blood will be discarded and would not be used, only the clear FF will be used.
* No flushing was used after oocyte aspiration in order not to interfere with the concentration of growth factors in the FF .

After explaining the procedure and taking informed consent from the patients:

2ml of clear follicular fluid will be injected in the uterine cavity to flush the endometrium through an IUI catheter after performing mock transfer in the study group.

While, in the control group, no flushing of the endometrial cavity with FF is done.

In both groups, embryo transfer will be carried out 2-3 days later according to the condition of the embryos and pregnancy test will be carried out 14 days later.

The protocol was approved by the review board at kasr el-Aini hospital; IVF center at Cairo university.

ELIGIBILITY:
Inclusion Criteria:

1. Maternal age ranges from 20-38 years.
2. Basal FSH < 10 mIU/ml.
3. BMI < 35 kg/m2.
4. Estradiol level > 1000 at the day of HCG administration.
5. Estradiol level < 4000 at the day of HCG administration.

Exclusion Criteria:

1. Presence of Endometriosis.
2. Presence of Hydrosalpinx.
3. Presence of vaginal infection.
4. Presence of galactorrhea.
5. Presence of hormonal disorders.
6. Severe male factor infertility:

   Sperm Count < one million. Marked malformation
7. history of recurrent abortion.

Ages: 20 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2011-12; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
pregnancy rate | 17 days
  The main outcome is the pregnancy rate in ICSI cycles after flushing the uterine cavity with follicular fluid after ovum pick-up in the study group and comparing it with the control group.

SECONDARY OUTCOMES:
Implantation rate | 17 days
  The secondary outcome is the implantation rate in ICSI cycles after flushing the uterine cavity with follicular fluid after ovum pick-up in the study group and comparing it with the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Nawara Mohamed Hashish, MD, Principal Investigator — Department of Obstetrics and Gynecology,Cairo University
Locations (1):
- Kasr El-Aini hospital, Cairo, Egypt